CLINICAL TRIAL: NCT04266691
Title: Molecular Metastasis in Lymph Nodes is Associated With Survival of Patients With Stage I NSCLC
Brief Title: Analysis of Driver Gene Mutation in Early Stage Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, zjszlyyad@126.com, Director of pathology, Zhejiang Cancer Hospital
Other Study IDs: LN-OMs
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Regional Lymph nodes; Molecular metastasis; Driver gene mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Driver gene mutation-positive: Screen the enrolled patients according to the admission criteria. The detection of lung cancer Polymerase Chain Reaction (PCR) panel kit in the hospital requires the use of tissue samples and the results show a driver gene mutation positive.
  Interventions: Other: nonIntervention
- Driver gene mutation-negative: Screen the enrolled patients according to the admission criteria. The detection of lung cancer Polymerase Chain Reaction (PCR) panel kit in the hospital requires the use of tissue samples and the results show a driver gene mutation negative.
  Interventions: Other: nonIntervention

INTERVENTIONS:
Other: nonIntervention — nonIntervention

SUMMARY:
Analysis of driver gene variation in early stage non-small cell lung cancer

DETAILED DESCRIPTION:
Fluorescence quantitative polymerase chain reaction (PCR) was used to detect the variation of driver gene in regional lymph nodes of early stage non-small cell lung cancer (NSCLC), and to analyze the relationship between the variation and disease recurrence and survival prognosis. evaluate the effect of the variation of driving gene in lymph nodes of early stage NSCLC on prognosis, identify the high-risk factors that promote the recurrence and metastasis of early stage tumor. so as to improve the diagnosis and treatment path of lung cancer, provide important pathological basis for the clinical diagnosis and treatment of early stage non-small cell lung cancer, enable patients to receive more accurate treatment, and improve their survival prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, 18 years of age or older
2. Histologically or cytologically proven diagnosis of early stage NSCLC
3. The lesion was completely resected by radical surgery
4. Able to get tumor tissue sample
5. Complete information of clinicopathological , survival, recurrence and metastasis can be obtained through follow-up

Exclusion Criteria:

1. Combine with other tumor type
2. The investigator judges the situation that may affect the clinical search process and results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically proven diagnosis of early stage NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Driver gene mutation frequency of early stage NSCLC | 2019
  Observe the driver gene mutation frequency in regional lymph nodes of early stage non-small cell lung cancer
Correlation of Clinicopathological characteristics and driver gene mutation in regional lymph nodes of early stage NSCLC | 2019
  Analyze the correlation between driver gene mutation and clinicopathological features in regional lymph nodes of early stage NSCLC
Correlation between driver gene mutation and survival prognosis in regional lymph nodes of early stage NSCLC | 2019
  Observe the correlation between driver gene mutation and survival prognosis in regional lymph nodes of early stage NSCLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian Y, Lai Q, Zheng Y, Ying L, Wang C, Jin J, Huang M, Wu Y, Li H, Zhang J, Su D. Oncogenic Alterations in Histologically Negative Lymph Nodes Are Associated with Prognosis of Patients with Stage I Lung Adenocarcinoma. Cancers (Basel). 2022 Feb 6;14(3):824. doi: 10.3390/cancers14030824. PMID 35159091